CLINICAL TRIAL: NCT06645470
Title: Muscle Quantity and Quality, With and Without Exercise, Combined With Anti-Obesity Medications
Brief Title: Muscle and Movement With Anti-Obesity Medications
Acronym: M3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Renee Rogers, Senior Scientist, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00160240; P20GM144269 (NIH)
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Obesity and Overweight
Keywords: exercise; weight loss; obesity medication; obesity; overweight
MeSH Terms: conditions — Obesity; Overweight; Motor Activity; Weight Loss | interventions — Resistance Training; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: 2-part design:
  (1) Randomized Pre-Post Parallel Design - 30 adults (18-<59 years) will be recruited that are newly prescribed an anti-obesity medication and randomize 10 to each of the intervention conditions.
  Randomized to:
  1. Standard Medical Care only,
  2. Standard Medical Care + aerobic training,
  3. Standard Medical Care + resistance training
  (2) Parallel longitudinal observational design - 10 older adults (>= 60 years) will be recruited that are newly prescribed an anti-obesity medication for observation.
  An additional subset of older adults taking an Anti-Obesity Medication (no exercise training).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Medical Care (Active Comparator): Standard Medical Care will continue to receive their regular standard clinical care during the 6-month intervention period of this study and will also receive brief contacts from the research staff at weeks 6, 12, and 18.
  Interventions: Other: Standard Medical Care (SMC); Behavioral: Monitoring Contacts; Other: Nutrition Education
- Standard Medical Care plus Aerobic Training (Experimental): Standard Medical Care plus Aerobic Training will continue to receive their regular standard clinical care during the 6-month intervention period of this study and will also receive supervised aerobic exercise in addition to brief contacts from the research staff at weeks 6, 12, and 18.
  Interventions: Other: Standard Medical Care (SMC); Behavioral: Monitoring Contacts; Behavioral: Aerobic Training; Other: Nutrition Education
- Standard Medical Care plus Resistance Training (Experimental): Standard Medical Care plus Resistance Training will continue to receive their regular standard clinical care during the 6-month intervention period of this study and will also receive supervised resistance exercise in addition to brief contacts from the research staff at weeks 6, 12, and 18.
  Interventions: Other: Standard Medical Care (SMC); Behavioral: Monitoring Contacts; Behavioral: Resistance Training; Other: Nutrition Education

INTERVENTIONS:
Other: Standard Medical Care (SMC) — Standard Medical Care will continue to receive their regular standard clinical care during the 6-month intervention period of this study.
Behavioral: Monitoring Contacts — Participants will receive contacts with the research staff at weeks 6, 12, and 18.
Behavioral: Aerobic Training — Aerobic Training will be supervised exercise. It will occur on 3 days per week and will progress to 50 minutes per session (150 minutes per week). The intensity of the exercise will progress from 60%±5% to 70%±5% of age-predicted maximal heart rate (if taking beta-blocker medication intensity will progress from a Rating of Perceived Exertion of 11-13 to 12-14 based on the 6-20 Borg scale). While walking will be the preferred mode of exercise, alternative forms of cardiovascular exercise (upright cycling, elliptical, etc.) are allowed to accommodate any physical limitations that may be present for a participant. Heart rate will be monitored throughout these exercise sessions.
  Arms: Standard Medical Care plus Aerobic Training
Behavioral: Resistance Training — Resistance Training will be supervised exercise. It will occur 3 days per week and includes 8 exercises performed in a prespecified order. Week 1-2 sessions focus on familiarization to acclimate the participant to the equipment, proper form, to establish initial weight (load) for training, and with performing multiple sets per day. For Weeks 3-8, participants will engage in 2 sets per exercise with the weight adjusted to elicit muscle fatigue in 8-12 repetitions per set. This progresses to 3 sets per exercise from Week 9 until the end of the intervention period. When 12 repetitions for a specific exercise can be achieved, the resistance will increase for that exercise at the next session. There is a 90 second rest period between each set of an exercise. Heart rate will be monitored throughout these exercise sessions.
  Arms: Standard Medical Care plus Resistance Training
Other: Nutrition Education — A single counseling session to discuss the dietary recommendations when taking an obesity medication.

SUMMARY:
The goal of this clinical trial is to learn about changes in body composition related to obesity medication use, and whether aerobic or resistance exercise training will impact these body composition changes. It will also provide information about whether aerobic or resistance exercise training has additional benefits on other health and fitness measurements. The main questions it aims to answer are:

* Is there a difference in the change in body composition (fat mass, lean mass, muscle mass, and bone content) between the standard medical care and the exercise conditions (aerobic training and resistance training)?
* Is there a difference in the change in body weight and BMI between the standard medical care and the exercise conditions (aerobic training and resistance training)?
* Is there a difference in the change in cardiorespiratory fitness between the standard medical care and the exercise conditions (aerobic training and resistance training)?
* Is there a difference in how much physical activity is completed between the standard medical care and the exercise conditions (aerobic training and resistance training)?
* Is there a difference in the change in physical function between the standard medical care and the exercise conditions (aerobic training and resistance training)?
* Is there a difference in the change in muscle strength between the standard medical care and the exercise conditions (aerobic training and resistance training)?
* Is there a difference in the change in resting blood pressure between the standard medical care and the exercise conditions (aerobic training and resistance training)?
* Is there a difference in the change in food intake between the standard medical care and the exercise conditions (aerobic training and resistance training)?
* Is there a difference in the change in health-related quality of life between the standard medical care and the exercise conditions (aerobic training and resistance training)?

Participants will:

* Participate in an intervention for a period of 6 months that involves being assigned to a no exercise/standard medical care condition, or a supervised exercise condition (aerobic training or resistance training).
* Visit the clinical before starting the study and at 6 months to complete study measurements of their body composition and other measurements to monitor their progress.
* Complete a brief monitoring session at weeks 6, 12, and 18 across the 6 months.
* Complete supervised exercise sessions at the research center 3x per week for 6 months (Participants in the exercise groups only: aerobic training or resistance training).

ELIGIBILITY:
Inclusion Criteria:

* Both males and females of all race/ethnic groups are eligible for participation in this study.
* Age: Randomized Study: Adults that are 18 to <60 years of age. Observational Study: Adults that are >60 years of age.
* Newly prescribed AOM (semaglutide, tirzepatide) for the treatment of obesity, approval for treatment (pharmacy, insurance, etc.), and the participant agreeing to start this treatment and continue treatment for at least 6 months (the participant will be recruited prior to this medication being initiated).
* Body mass index (BMI) of >27.0 kg/m2 with at least one weight-related complication (hypertension, dyslipidemia, obstructive sleep apnea, or cardiovascular disease) provided it this does not compromise the ability to safely complete the screening or outcome measures or to engage in the prescribed exercise interventions), or >30 kg/m2 without weight-related complications. Enrollment will not be limited based on an upper BMI level provided that the participant meets the other eligibility requirements. However, weight or size limits of the dual-energy x-ray absorptiometry (DXA) system that is used to assess body composition must not be exceeded.
* Ability to provide informed consent prior to participation in this study.
* Clearance from the study physician for meeting all eligibility criteria for this study.

Exclusion Criteria:

* Type 2 diabetes.
* Report moderate-to-vigorous exercise for >60 min/week, and >1 day of structured cardiovascular or resistance exercise over the past 3 months.
* Report sustained weight loss of >3% in the past 3 months.
* History of metabolic/bariatric surgery.
* Females who are pregnant, pregnant within the past 6 months, or reporting a planned pregnancy during the study period.
* Report a current medical condition or treatment for a medical condition that could affect body weight or contradict engagement in any aspect of the outcome measures or interventions.
* History of muscle conditions that may impact the quality of muscle or response to the study interventions (e.g., myopathy, muscular dystrophy, rhabdomyolysis, etc.).
* Current congestive heart failure, angina, uncontrolled arrhythmia, symptoms indicative of an increased acute risk for a cardiovascular event, prior myocardial infarction or history of cardiomyopathy, coronary artery bypass grafting or angioplasty, conditions requiring chronic anticoagulation (i.e., recent or recurrent DVT).
* Resting systolic blood pressure of >160 mmHg or resting diastolic blood pressure of >100 mmHg. If medicated for blood pressure control, the medication dose needs to be stable for >6 months.
* Eating disorders that would contraindicate weight loss or physical activity.
* Alcohol or substance abuse.
* Current psychological condition that is untreated, hospitalization for a psychological condition within the past 12 months, or not being on a stable dose of treatment for at least 6 months.
* Report plans to relocate to a location not accessible to the study site or having employment, personal, or travel commitments that prohibit attendance at scheduled intervention sessions or assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lean Body Mass | 0 and 6 months
  Lean body mass (kg) will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).

SECONDARY OUTCOMES:
Body Fat Mass | 0 and 6 months
  Body fat mass (kg) will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Percent Body Fat | 0 and 6 months
  Percent body fat will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Body Weight | 0 and 6 months; 6, 12, 18 weeks
  Body weight will be assessed in duplicate using a calibrated digital scale to the nearest 0.1 kg.
Body Height | 0 and 6 months; 6, 12, and 18 weeks
  Body height will be assessed in duplicate using a wall mounted stadiometer to the nearest 0.1 cm.
Body Mass Index | 0 and 6 months; 6, 12, 18 weeks
  Measurements of weight and height will be used to compute BMI (kg/m2).
Bone Mineral Content | o and 6 months
  Bone mineral content (grams) will be assessed using a total body scan from dual-energy x-ray absorptiometry (DXA).
Muscle Mass | 0 and 6 months
  Muscle mass will be assessed using the deuterated creatine (D3Cr) dilution method. A 30mg capsule of D3Cr is ingested and 48-72 hrs later, a fasting urine sample is provided for analysis.
Muscular Strength | 0 and 6 months
  Muscular strength will be assessed using isometric leg extension on a Biodex.
Muscular Strength | 0 and 6 months
  Muscular strength will be assessed using grip strength with a hand grip dynamometer.
Physical Function | 0 and 6 months
  Physical Function will be assessed using the Short Physical Performance Battery (SPPB) that includes balance, gait speed, and chair stands. A composite score with a range from 0 to 12 (no units) of these measures is used. A higher score represents better physical functioning.
Cardiorespiratory Fitness | 0 and 6 months
  Cardiorespiratory fitness will be represented as milliliters of oxygen consumed per kilogram of body weight per minute (ml/kg/min) measured with a metabolic cart during a submaximal graded exercise test that is terminated when the participant achieves 85% of age-predicted maximal heart rate.
Cardiorespiratory Fitness | 0 and 6 months
  Cardiorespiratory fitness will be represented as total liters of oxygen consumed per minute (L/min) measured with a metabolic cart during a submaximal graded exercise test that is terminated when the participant achieves 85% of age-predicted maximal heart rate.
Cardiorespiratory Fitness | 0 and 6 months
  Cardiorespiratory fitness will be the duration measured in minutes to achieve 85% of age-predicted maximal heart rate during a submaximal graded exercise test performed on a treadmill.
Resting Blood Pressure | 0 and 6 months; 6, 12, and 18 weeks
  Resting seated blood pressure, both systolic and diastolic (mmHg), will be assessed using an automated system.
Energy Intake (Dietary Intake) | 0 and 6 months
  Energy Intake (Dietary Intake) expressed as kilocalories eaten per day (kcal/day) will be measured using the Diet History Questionnaire (DHQ) developed by NCI. A higher score represents more calories eaten.
Physical Activity | 0 and 6 months
  Physical activity is measured by the Global Physical Activity Questionnaire (GPAQ). This assesses time spent in recreational, occupational, household, and transportation physical activities and is represented as minutes per week. Higher minutes per week indicate greater physical activity participation. The range is 0 to 10,080 minutes per week.
Health-Related Quality of Life | 0 and 6 months
  Health-Related Quality of Life will be measured with a 36-item questionnaire (RAND 36-Item Health Survey) that includes 8 subscales of vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health or emotional wellbeing. All items are scored so that a high score defines a more favorable health state. The range of the final score for each subscale is 0-100.

OTHER OUTCOMES:
Demographic Characteristics | 0 months
  Demographic Characteristics will be assessed using a survey.
Lifestyle and Health History | 0 months
  A questionnaire developed specifically for this study that is conducted as an interview will be used to assess lifestyle and health factors to describe the sample for this study. The score is either "yes" or "no" identifying the presences of a lifestyle or health factor.
Medication History | 0 and 6 months; 6, 12, and 18 weeks
  A questionnaire developed specifically for this study will be used to assessment medication history. The data collected include the type of medication, dose of medication, and frequency that the medication is taken, and what condition the medication is indicated to treat.
Adverse and Serious Adverse Events | 0 and 6 months; 6, 12, and 18 weeks
  Participants will be queried using a survey developed specifically for this study will be used to assess for adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Renee J. Rogers, Ph.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The summary data for each of the study outcomes and other additional demographic characteristics will be made available. The Study Protocol (which includes the statistical analysis plan), Manual of Procedures, Data Collection Forms, and a Data Dictionary to explain the data variables will be provided.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available no later than the time of an associated publication of study outcomes or at the end of the performance period, whichever comes first. The data provided to the repository will be available indefinitely while that repository continues to exist.
Access Criteria: The information included with the IPD will be made available to appropriate individuals only after the requester confirms their willingness to comply with an appropriate "Data Use Agreement" that complies with NIH policies, the policies of the institution where the study has been conducted, and the elements of informed consent.

REFERENCES:
- [Derived] Jakicic JM, Rogers RJ. The Role of Exercise in the Contemporary Era of Obesity Management Medications. Curr Sports Med Rep. 2025 Aug 1;24(8):240-245. doi: 10.1249/JSR.0000000000001272. PMID 40758789